CLINICAL TRIAL: NCT00280761
Title: A Biologic Study of Global Gene Expression, NF-Kappa B and p53 in Adenocarcinoma of the Rectum.
Brief Title: Biomarkers in Patients With Rectal Cancer Undergoing Chemotherapy and Radiation Therapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 0216; P30CA016086 (NIH); CDR0000561688 (Other: PDQ number)
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; recurrent rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adenocarcinoma of the Rectum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Single Arm Trial
  Interventions: Drug: capecitabine; Drug: 5-fluorouracil; Procedure: Surgical Resection; Radiation: Radiation therapy

INTERVENTIONS:
Drug: capecitabine — Capecitabine administration (where deemed appropriate by the treating medical oncologist) will commence on the second day of radiotherapy after the 24-hour biopsy has been performed. Dosing will be per current standard of care at the discretion of the treating Medical, Radiation and Surgical Oncologist
  Other Names: Xeloda
Drug: 5-fluorouracil — Administration of 5-fluorouracil (where deemed appropriate by the treating medical oncologist) will commence on the second day of radiotherapy after the 24-hour biopsy has been performed. Dosing and dose modification will be per current standard of care at the discretion of the treating Medical, Radiation and Surgical Oncologist.
  Other Names: 5-FU
Procedure: Surgical Resection — Surgery will occur approximately 2-6 weeks after chemoradiation depending on clinical factors (i.e. resectability, presence or absence of metastatic disease).
Radiation: Radiation therapy — Dosing and dose modification will be per current standard of care at the discretion of the treating Radiation Oncologist.
  Other Names: EBRT - External Beam Radiation Therapy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand how patients respond to treatment.

PURPOSE: This clinical trial is studying biomarkers in patients with rectal cancer undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Observe whether NF-kappa B is activated in response to treatment with external beam radiotherapy.
* Correlate NF-kappa B pathway activation (presumed to be anti-apoptotic in nature) with therapeutic outcomes (as measured by rate of pathologic complete response or downstaging by endoscopic ultrasound [EUS]).

Secondary

* Study downstream events induced by NF-kappa B activation.
* Determine global gene expression profiles at baseline and during chemoradiotherapy.
* Correlate changes in gene expression (compared with the baseline gene expression pattern) induced by a single dose of external beam radiotherapy with patient outcomes (as measured by pathologic response rate or downstaging by EUS).
* Study downstream events related to activation of p53 in response to treatment with radiotherapy.
* Correlate p53 pathway-mediated events with clinical outcomes.

OUTLINE: Patients receive fluorouracil or capecitabine and undergo radiotherapy and surgery per standard care.

Patients undergo tumor pinch biopsies at baseline and on days 1 and 2 of chemoradiotherapy. At the time of final surgical resection, a portion of the remaining rectal tumor will be liquid nitrogen banked. Patients not deemed surgical candidates are evaluated by transrectal ultrasound 6-8 weeks after completion of chemoradiotherapy to assess ultrasound response (downstaging versus no downstaging).

Tumor tissue samples are analyzed for NF-kappa B pathway activation; downstream events induced by NF-kappa B activation; changes in global gene expression; p53 function; apoptosis; and mRNA expression. Laboratory techniques used include tissue microarray, ELISA, RNase protection assay, fluorescence semi-quantitative PCR, TUNEL, IHC, and cDNA microarray analysis.

If normal tissue from biopsies is not available, whole blood may be collected at any point while patient remains on study for correlative analysis or research related to rectal cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have rectal or sigmoid-rectal junction adenocarcinoma confirmed by sigmoidoscopy and pathologic diagnosis of biopsy sample

  * Inferior margin of the tumor less than 15 cm from anal verge by rigid sigmoidoscopy or below the level of S1-2 at surgery
* Candidate for chemotherapy and radiotherapy, as defined by any of the following:

  * Tumor staged as T3 or N1-2 by rectal sonography
  * Tumor occupying > 40% of circumference of rectum
  * Tumor fixed to extra colonic structures as determined by digital rectal examination
  * Tumor < 5 cm from sphincter mechanism
  * Patient has inoperable disease and is being treated for palliation
  * Pelvic or anastomotic recurrences of previously resected rectal cancer
* Planning to undergo chemotherapy and radiotherapy
* No sigmoid carcinoma (carcinoma proximal to the pelvic peritoneal reflection)

PATIENT CHARACTERISTICS:

* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (male, female, any ethnic background) with rectal (inferior margin of the tumor less than 15cms from anal verge by rigid sigmoidoscopy or below the level of S1-2 at operation) or sigmoid-rectal junction carcinomas confirmed by sigmoidoscopy and pathologic diagnosis of biopsy sample.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2003-12; Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Activation of NF-kappa B in response to treatment with external beam radiotherapy | 6-8 weeks after chemoradiation
Correlation of NF-kappa B pathway activation with therapeutic outcomes | 6-8 weeks after chemoradiation

SECONDARY OUTCOMES:
Downstream events induced by NF-kappa B activation | 12 months
Global gene expression profiles at baseline and during chemoradiotherapy | prior to chemoradiation and 72 days post chemoradiation
Correlation of changes in gene expression with patient outcomes | 72 days post chemoradiation
Downstream events related to activation of p53 in response to treatment with radiotherapy | 72 post radiotherapy
Correlation of p53 pathway-mediated events with clinical outcomes | 72 days post chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sanoff, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: web address for UNC Lineberger Comprehensive Cancer Center — http://www.unclineberger.org/
- See also: web address for the National Cancer Institute (NCI) — http://www.cancer.gov/